CLINICAL TRIAL: NCT05257343
Title: Assessment of the Efficacy of a Low-Dose Iron Supplement in Restoring Iron Levels to Normal Range Without Promoting Constipation or Adverse Gastrointestinal Effects Among Healthy Premenopausal Women With Iron Deficiency Without Anemia
Brief Title: Efficacy of a Low Dose, Oral, Liquid Iron Supplement on Restoring Inadequate Blood Iron to Normal Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MF121521
Record Dates: First submitted 2022-02-04; First posted 2022-02-25 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: Iron Deficiency; Iron Supplementation; Premenopausal Women; Ferritin; Hematology
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel, placebo-controlled, 8-week intervention clinical study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily dose (10 mL) of a visually identical liquid placebo supplement to be ingested on an empty stomach no sooner than 3 hours after consuming a meal.
  Interventions: Dietary Supplement: Liquid Placebo Supplementation
- Blood Builder Treatment (Experimental): Daily dose (10 mL) of liquid iron supplement (Blood Builder®) formulation to be ingested on an empty stomach no sooner than 3 hours after consuming a meal.
  Interventions: Dietary Supplement: Liquid Iron Supplement (Blood Builder ®)

INTERVENTIONS:
Dietary Supplement: Liquid Placebo Supplementation — 8-weeks of supplementing with a visually identical liquid placebo supplement.
  Arms: Placebo
Dietary Supplement: Liquid Iron Supplement (Blood Builder ®) — 8-weeks of supplementing with a liquid iron supplement (Blood Builder ®)
  Arms: Blood Builder Treatment

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 8-week intervention clinical study assessing the safety and efficacy of a new low-dose liquid iron supplement in restoring iron levels to normal ranges without promoting constipating side-effects among healthy premenopausal women with non-anemic iron deficiency. The primary outcomes will be an Iron Panel of Serum Iron, Ferritin, Total iron-binding capacity, Transferrin saturation, Complete Blood Count, and high sensitivity - C-Reactive Protein. Secondary outcomes will be surveys on gastrointestinal distress/discomfort and well-being. Adverse events will also be reported.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 8-week intervention clinical study assessing the safety and efficacy of a new low-dose liquid iron supplement in restoring iron levels to normal ranges without promoting constipating side-effects among healthy premenopausal women with non-anemic iron deficiency.

A total of 82 premenopausal female subjects over the age of 18 years old are planned for this study. Enrolled subjects will be assigned a unique study number in the 100 series as the subject ID for the study to maintain anonymity. The subject ID will be assigned in sequential order starting with 101 (i.e., 101, 102, 103, etc). After signing the informed consent document, enrolled subjects will be screened, and qualifying subjects will be randomly assigned to one of two groups (Group A or Group B) depending on the treatment (liquid iron supplement or placebo). Following random assignment, subjects will revisit the laboratory to complete baseline testing for primary, secondary, and exploratory outcomes. After 4 weeks of daily supplementation of their respective randomly assigned condition, subjects return to the laboratory for reassessment of secondary outcomes. The last laboratory visit will occur following 8 weeks of daily supplementation in which subjects will be reassessed on all outcomes in a manner identical to baseline.

GROUPS:

* Group A: Single-dose containing 10 mL of a liquid iron formulation to be ingested once a day on an empty stomach no sooner than 3 hours after consuming a meal.
* Group B: Single-dose containing 10 mL of the placebo formulation to be ingested once a day on an empty stomach no sooner than 3 hours after consuming a meal.

VISITS:

* Visit 1: Study enrollment and eligibility screening. Written informed consent will be obtained to confirm study enrollment prior to eligibility screening.
* Visit 2: Baseline assessment
* Visit 3: Reassess secondary variables only
* Visit 4: Reassess all measurements for final post-testing and end of study (EOS).

For laboratory visits requiring blood donation (visits 1, 2, and 4), subjects will arrive at the laboratory following an overnight fast (≥ 10 hours) and undergo standard sterile venipuncture techniques by a certified phlebotomist. Blood samples, approximately 10mL in volume, will be collected into a marble top (gel-barrier) tube interiorly coated with silicone. Following collection, samples will be inverted 4-6 times then stored upright at room temperature in a test tube holder for approximately 30 minutes to promote coagulation; thereafter, samples will be centrifuged for serum separation. The resulting serum aliquot will be immediately stored at -80°C until further analysis of blood chemistry variables.

For questionnaire assessments (Patient assessment of constipation - symptoms, functional bowel index, Gastrointestinal symptom rating scale, and abbreviated Profile of Mood States), subjects will complete the questionnaires in isolation in a quiet room isolated to avoid bystander influence. For visit 3, subjects are not required to be fasted. All study visits will be conducted at the same time of day (± 1 hour).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects > 18 years old
* Premenopausal (experiencing regular menstrual cycles)
* Hemoglobin > 11g/dL
* Serum ferritin < 70 ng/mL
* hs-CRP < 3 mg/L
* BMI 18 - 29.9 kg/m2
* No intake of dietary supplements containing iron 30 days prior to enrollment
* Willing and able to give written informed consent
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the schedule visit(s) and study requirements.

Exclusion Criteria:

* Currently taking (within the past 14 days) dietary supplements including, vitamins (any), minerals, protein shakes, vitamin water, other supplements
* History of gastrointestinal disorders that could lead to uncertain absorption of the study supplements, (i.e., inflammatory bowel disease, ulcerative colitis, Crohn's disease, colostomy, or eating disorder)
* History or current malignancy
* Receiving chemotherapy agents or radiation treatments
* Prior health issues showing high CRP or other inflammatory markers
* Pregnancy or has breast fed within 3 months prior to enrollment
* BMI <18 or >25 kg/m2
* Diagnosis of a terminal illness
* Use of prescription medications that impact digestion (i.e., proton pump inhibitor medications, other)
* History of alcohol abuse
* History or current drug abuse
* History or current cigarette smoke (including vaping) within the past 14 days from the screening visit
* Insulin-dependent diabetes and/or metformin use
* Chronic kidney or liver disease
* Anemia
* Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, hepatitis B/C, HIV, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years, or other, which in the opinion of the investigator, such condition might be aggravated as a result of treatment
* The investigator feels that for any reason the subject is not eligible to participate in the study
* Use within 24 hours preceding enrollment of ibuprofen, acetaminophen, any other analgesics, anti-inflammatory products, or any products including herbals and supplements that could interfere with the clinical assessments of this study (other than drugs used for anesthesia)
* History of uncontrolled cardiovascular disease (i.e., myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* History, or current bleeding disorders (i.e., hemophilia or von Willebrand disease), or anticipated treatment with prescription anticoagulants
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* A family member of the investigator or an employee of the investigator
* Participation in any other investigational study within 30 days prior to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Serum Iron | Week 0 and Week 8
  Changes in Iron in fasted serum blood samples.
Serum Ferritin | Week 0 and Week 8
  Changes in Ferritin in fasted serum blood samples.
Total Iron-Binding Capacity (TIBC) | Week 0 and Week 8
  Changes in TIBC in fasted serum blood samples.
Transferrin Saturation (tSAT) | Week 0 and Week 8
  Changes in tSAT in fasted serum blood samples.
Complete Blood Count (CBC) | Week 0 and Week 8
  Changes in complete blood count with differential will be assessed via fasted serum blood samples
High Sensitivity C-Reactive Protein (hs-CRP) | Week 0 and Week 8
  Changes in hs-CRP in fasted serum blood samples.

SECONDARY OUTCOMES:
Patient Assessment of Constipation - Symptoms Questionnaire | Week 0, Week 4, and week 8
  Changes assessed by administering the Patient Assessment of Constipation - Symptoms questionnaire for subjective assessment of constipation symptoms. Each question is answered from 0 (no symptoms at all) to 4 (severe symptoms). The lower the mean score, the less severe the symptoms. The higher the mean score, the more severe the symptoms.
Functional Bowel Index | Week 0, Week 4, and week 8
  Changes assessed by administering the Functional Bowel Index for subjective assessment of bowel movements. A 3 item questionnaire scored from 0-100 with higher scores indicating greater severity and scores higher than 28.8 points indicating constipation.
Gastrointestinal symptom rating scale | Week 0, Week 4, and week 8
  Changes assessed by administering the Gastrointestinal Symptom Rating Scale for subjective assessment of gastrointestinal symptoms and their severity. It is a 15-item questionnaire designed to assess the symptoms associated with common GI disorders. It has 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). Subscale scores range from 1 to 7 and higher scores represent more discomfort, and lower scores represent less or even no discomfort.
Abbreviated Profile of Mood States | Week 0 and Week 8
  Changes assessed in the abbreviated profile of mood states for subjective assessment of the subject's mood and overall well-being. It is a 40 point scale, divided into 7 different subscales, with a 5 point Likert scale, ranging from 0 (not at all) to 4 (Extremely) of how a subject feels in response to that particular feeling. The following equation is used to determine the overall score: Total Mood Disturbance = [Tension+Depression+Anger+Fatigue+Confusion] - [Vigor+Esteem Related Affect]. A lower score indicates overall better mood, while a lower score indicates worse overall mood.
Adverse Events | Week 0, Week 4, and Week 8
  Defined as participants self-reported adverse effects. Items that will be surveyed are headache, dizziness, nausea, vomiting, indigestion, blurred vision, lethargy, swelling, itching, chest pain, heart palpitations, difficulty breathing, lethargy, and muscle cramps.

OTHER OUTCOMES:
Body Composition via Body Fat Percentage | Week 0 and Week 8
  Changes assessed in body fat percentage via Dual X-Ray Absorptiometry.
Bone Mineral Density | Week 0 and Week 8
  Changes assessed in bone mineral density in grams via Dual X-Ray Absorptiometry.

CONTACTS AND LOCATIONS:
Locations (1):
- The Applied Science and Performance Institute, Tampa, Florida, United States